CLINICAL TRIAL: NCT00144352
Title: The in-Vivo Response of P. Falciparum to Antimalarial Treatment in HIV-Infected and HIV-Uninfected Individuals-a 28 Day Efficacy Trial Involving HIV+ and HIV- Adults.
Brief Title: In-Vivo Response of P. Falciparum to Antimalarial Treatment in HIV-Infected and HIV-Uninfected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCID-3537; UR6/CCU018970-02-2; SCC#644
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Malaria; HIV; AIDS
Keywords: Malaria; HIV; AIDS; drug efficacy; Kenya; Africa; Sulfadoxine pyirmethamine; fansidar
MeSH Terms: conditions — Malaria; Acquired Immunodeficiency Syndrome | interventions — fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine

SUMMARY:
Plasmodium falciparum malaria and HIV are among the most important infectious diseases in sub-Saharan Africa. Approximately two-thirds of the estimated 35 million HIV infected persons live in sub-Saharan Africa. Of the 300-500 million annual cases of malaria infection occurring worldwide, about 90% of P. falciparum infections occur in sub-Saharan Africa, resulting in approximately 1 million deaths, mostly in children under five years of age. It is clear that HIV and malaria are responsible for substantial disease, suffering, and an enormous economic burden on the people who can least afford it. Although a study in 1993 in Tanzania showed significantly higher prevalence of malaria infections in HIV-positive compared to HIV negative adults, until recently there have been few studies showing any association between the two infections.

We conducted a study to measure the efficacy of the then-first line antimalarial drug (sulfadoxine-pyrimethamine) among patients in three study arms: those who were HIV negative, those who were HIV infected with CD4 cell counts < 200, and among HIV infected patients with CD4 cell counts >= 200. Our hypothesis is that patients with HIV infection and low CD4 cell count will not respond to antimalarial therapy as well as patients who are HIV infected with higher CD4 cell counts or who are HIV negative.

DETAILED DESCRIPTION:
The study was conducted at Siaya District Hospital, in Nyanza Province, Kenya. Non-pregnant adults who provided consent to participate, who were found to have pure Plasmodium falciparum malaria parasitemia with at least 500 asexual parasites per microliter, and who agreed to undergo HIV counseling and testing were eligible for participation. Clients were then followed with repeat physical examinations and blood smears on day 1,2,3,4,7,14,21 and 28 and any non-scheduled day when they were sick. Those that failed therapy were treated with quinine to clear parasitemia. Samples were also taken to measure reinfection vs. recrudescence, pharmacokinetics, and antifolate resistance markers.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older, not pregnant. Are able to make all follow-up visits. Are able to understand and give informed consent. Have a history of fever in past 24hrs or current axillary temperature of ³ 37.5C.

Have an unmixed infection with P. falciparum of at least 500 asexual parasites/mm3 as determined by microscopic examination of thick and/or thin peripheral blood smears.

Do not have any evidence of severe or complicated malaria (e.g., cerebral malaria, Hb < 5 g/dL, signs and symptoms of congestive heart failure) that would require hospitalisation for treatment.

Have no reported allergy to sulfa drugs. Agree to HIV testing and receiving the results.

Exclusion Criteria:

Less than 18 yrs old. Pregnant. History of allergic reactions to sulfa drugs. Have severe or complicated malaria. No history of fever. Plan to leave Siaya in next month. Do not agree to HIV testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540
Dates: Start 2002-09; Study Completion 2004-07

PRIMARY OUTCOMES:
Drug failure

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Shah, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- CDC KEMRI Research Institute, Kisumu, Kenya